CLINICAL TRIAL: NCT01470066
Title: Clinical Usefulness and Prognostic Significance of Interim 18F-FDG PET/CT for the Treatment of Peripheral T Cell Lymphomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other)
Other Study IDs: PET2005-01
Record Dates: First submitted 2011-11-03; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2005-09

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T cell lymphomas; interim PET/CT; prognosis; Positron-emission tomography/Computerized tomography
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although interim 18F-fluoro-2-deoxy-D-glucose-positron emission tomography (FDG-PET)/computerized tomography (CT) scan has emerged as a powerful prognostic tool in predicting treatment outcome in Hodgkin's lymphoma (HL) and diffuse large B cell lymphoma (DLBCL), the positive predictive value (PPV) of interim PET/CT scanning has not been determined in patients with peripheral T cell lymphoma (PTCL). The sequential interim PET/CT will be prospectively investigated to determine whether it provided additional prognostic information and could be a positive predictable value for the treatment of PTCL.

DETAILED DESCRIPTION:
1. Treatment protocol

   * Patients with limited-stage (stage I/II) are treated with CHOP/CHOP-like chemotherapy [cyclophosphamide 750 mg/m2 i.v. on D1, vincristine 1.4 mg/m2 i.v. on D1, doxorubicin 50 mg/m2 i.v. on D1, and prednisolone 60 mg/m2 p.o. on D1-5] in standard doses every three weeks and three to four cycles of CHOP/CHOP-like chemotherapy followed by involved field radiation therapy (IFRT, 30 Gy). Patients with advanced-stage (stage III/IV) are treated with eight cycles of primary chemotherapy and patients greater than 65 years and/or those with a frail general condition were treated with only six cycles of primary chemotherapy if they achieved a complete response (CR) for the interim response.
2. Response evaluation based on three parameters of visual, standard uptake value(SUV)-based and metabolic tumor volume (MTV)-based assessments

   * We firstly classify patients with five-point scale (5-PS) by the interim PET/CT analysis based on the Deauville criteria12: 1, No uptake; 2, uptake ≤ mediastinum; 3, uptake > mediastinum but ≤ liver; 4, uptake moderately increased compared to the liver uptake at any site; 5, markedly increased uptake compared to the liver at any site and new sites or/and new sites of disease. Interim PET/CT image are graded as negative or positive by comparison of initial PET/CT and grade 1-3 considered as negative and grade 4-5 considered for positive.19 This grading process is independent of the size of the residual tumor.

   Secondly, we classify the patients with the quantitative analysis of 18F-FDG uptake changes based on the percentage of SUVmax reduction between initial and interim PET/CT. On axial, coronal, or sagittal coregistered PET/CT slices, simple circular regions of interest (ROIs) were placed so as to cover the lesion or background. SUV measurements are corrected for body weight according to the following standard formula: Mean ROI activity (MBq/ml)
   * [Injected dose (MBq)/Body weight (kg)].20 For each PET dataset, the maximum SUV (SUVmax) is defined as the highest SUV among all hypermetabolic tumor foci. SUVmax reduction rate (ΔSUVmax) is calculated as following:

   ΔSUVmax (%) = 100 x [SUVmax (initial) - SUVmax (interim)]/SUVmax (initial)

   If all lesions had disappeared on interim PET, ROI were drawn in the same area on interim PET as on baseline PET.

   We finally classify the patients with the quantitative analysis of metabolic volume changes based on the percentage of MTV reduction (ΔMTV) between initial and interim PET/CT. To define the exact tumor margins around the target lesions, SUV2.5 is used as following previous reports, which means that the tumor volume area in PET/CT is delineated by a circle encompassing regions with SUV cutoff value of 2.5.16,21 The MTV2.5 is measured using AW Volume ShareTM workstation (GE Healthcare) on the fused PET/CT images.17 AW Volume ShareTM allows automatic registration and fusion between two volumetric acquisitions, which come from different acquisition modalities. The active MTV2.5 are measured in a 3-D manner by selecting volume of interest (VOI) on the axial image, and the size of VOI is manually regulated on the corresponding coronal and sagittal images to include entire active tumors in the VOI. The SUVmax and the sum of the tumor volumes in all hypermetabolic tumor foci were computed automatically by the program. The MTV2.5 reduction rate (ΔMTV2.5) is calculated as same formula as SUVmax reduction rate.
3. The response assessments of interim PET/CT scans

   * will be assessed based on the combination with three parameters of the Deauville five-point scale (5-PS), the reduction rate of maximal standardized uptake value (ΔSUVmax), and the reduction rate of metabolic tumor volume (ΔMTV2.5) in PTCLs

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Histologically proven PTCLs except primary cutaneous/subcutaneous panniculitis
3. ECOG performance status ≤ 2
4. Patients who are available to be performed PET/CT at diagnosis
5. No severe concomitant disease

Exclusion Criteria:

1. Patients who did not undergo PET/CT scans at diagnosis
2. Patients who have a primary CNS lymphoma
3. Patients who have a HIV or HTLV-1
4. Patients who could not receive primary chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is the observational study for the response assessments on interim PET/CT during the treatment of peripheral T cell lymphomas. Thus, first analysis of clinical data will be performed at the time of 80 patients enrolled or after a median follow-up of more than 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2004-08; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From the treatment start time to the first recording of disease progression or death from any cause, which assessed up to 24 months.
  Patients whose disease did not progress would be censored using the date at which they were last known to show no progress.

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

REFERENCES:
- [Derived] Jung SH, Ahn JS, Kim YK, Kweon SS, Min JJ, Bom HS, Kim HJ, Chae YS, Moon JH, Sohn SK, Lee SW, Byun BH, Do YR, Lee JJ, Yang DH. Prognostic significance of interim PET/CT based on visual, SUV-based, and MTV-based assessment in the treatment of peripheral T-cell lymphoma. BMC Cancer. 2015 Mar 28;15:198. doi: 10.1186/s12885-015-1193-1. PMID 25879747